CLINICAL TRIAL: NCT01830621
Title: A Phase III Randomized Study of BBI608 and Best Supportive Care Versus Placebo and Best Supportive Care in Patients With Pretreated Advanced Colorectal Carcinoma
Brief Title: BBI608 and Best Supportive Care vs Placebo and Best Supportive Care in Pretreated Advanced Colorectal Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CO23
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — napabucasin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BBI608 (Active Comparator): BBI608 480 mg two times daily (960 mg total daily dose)+ Best Supportive Care
  Interventions: Drug: BBI608; Other: Best Supportive Care
- Placebo (Placebo Comparator): Placebo two times daily + Best Supportive Care
  Interventions: Drug: Placebo; Other: Best Supportive Care

INTERVENTIONS:
Drug: BBI608
  Arms: BBI608
Drug: Placebo
  Arms: Placebo
Other: Best Supportive Care

SUMMARY:
The purpose of this study is to find out whether it is better to receive a new drug, BBI608, or better to receive no further treatment for colon or rectal cancer. To do this, half of the patients in this study will get BBI608 and the other half will receive a placebo (a substance that is designed not to do anything).

DETAILED DESCRIPTION:
This research is being done because currently there are no approved remaining effective treatments for colon or rectal cancer.

The purpose of this study is to compare the effects on colon cancer of a new drug, BBI608, and best supportive care (BSC) compared to BSC alone.

BBI608 has been shown to shrink tumours in animals and has been studied in a few people and seems promising, but it is not clear if it can offer better results than the usual care which is best supportive care alone.

The standard or usual treatment for this disease is treatment with drugs and other treatments that may help to make a patient feel better or may improve their quality of life. This treatment is known as "best supportive care" (BSC). Although patients with best supportive care can feel better for some months, the cancer usually continues to grow.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced colorectal cancer that is unresectable.
* Received a prior thymidylate synthase inhibitor (e.g. 5-fluorouracil (5-FU), capecitabine, raltitrexed, UFT) for metastatic disease or as adjuvant therapy.
* Received and failed an irinotecan containing regimen (i.e. single-agent or in combination) for treatment of metastatic disease, OR relapsed within 6 months of completion of an irinotecan-containing adjuvant therapy, OR have documented unsuitability for an irinotecan-containing regimen.
* Received and failed an oxaliplatin-containing regimen for treatment of metastatic disease, OR relapsed within 6 months of completion of an oxaliplatin-containing adjuvant therapy OR have documented unsuitability for an oxaliplatin-containing regimen.
* For patients with colorectal cancer that is K-ras wild type: Received and failed a cetuximab or panitumumab-containing regimen (i.e. single-agent or in combination) for treatment of metastatic disease OR have documented unsuitability for a cetuximab or panitumumab-containing regimen
* The only remaining standard available therapy as recommended by the Investigator is best supportive care.
* Must have presence of measurable disease as defined by Response Evaluation Criteria in Solid Tumours (RECIST 1.1).
* Imaging investigations including CT/MRI of chest/abdomen/pelvis or other scans as necessary to document all sites of disease done within 14 days prior to randomization.
* Must have an ECOG Performance Status of 0 or 1.
* Must be ≥ 18 years of age.
* For male or female patient of child producing potential: Must agree to use contraception or take measures to avoid pregnancy during the study and for 30 days after the last Protocol treatment dose.
* Women of child bearing potential (WOCBP) must have a negative serum or urine pregnancy test within 72 hours prior to randomization.
* Must have alanine transaminase (ALT) ≤ 3 × institutional upper limit of normal (ULN) [≤ 5 × ULN in presence of liver metastases] within 14 days prior to randomization.
* Must have hemoglobin (Hgb) ≥ 80 g/L within 14 days prior to randomization.
* Must have total bilirubin ≤ 1.5 × institutional ULN [≤ 2.0 x ULN in presence of liver metastases] within 14 days prior to randomization.
* Must have creatinine ≤ 1.5 × institutional ULN or Creatinine Clearance > 50 ml/min within 14 days prior to randomization.
* Must have absolute neutrophil count ≥ 1.5 x 109/L within 14 days prior to randomization.
* Must have platelet count ≥ 75 x 109/L within 14 days prior to randomization.
* Other biochemistry which must be done within 14 days prior to randomization includes lactate dehydrogenase (LDH) and alkaline phosphatase.
* Patient must consent to provision of, and investigator(s) must confirm access to and agree to submit at the request of the NCIC CTG Central Tumour Bank, a representative formalin fixed paraffin block of tumour tissue in order that the specific correlative marker assays may be conducted.
* Patient must consent to provision of a sample of blood in order that the specific correlative marker assays may be conducted.
* Patient is able (i.e. sufficiently fluent) and willing to complete the Quality of Life and Health Utilities questionnaires in one of the validated languages for the questionnaires.
* Patients must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating centre. This implies there must be reasonable geographical limits placed on patients being considered for this trial.
* Protocol treatment is to begin within 2 working days of patient randomization.
* The patient is not receiving therapy in a concurrent clinical study and the patient agrees not to participate in other clinical studies during their participation in this trial while on study treatment.

Exclusion Criteria:

* Anti-cancer chemotherapy or biologic therapy within the lesser of i) 21 days, or ii) the usual cycle length of the regimen (e.g. 14 days for FOLFOX), prior to the first planned dose of BBI608/placebo. An exception is made for capecitabine and regorafenib, where a minimum of 10 days since last dose must be observed prior to the first planned dose of BBI608/placebo.
* Radiotherapy, immunotherapy, or investigational agents within four weeks of first planned dose of BBI608/placebo, with the exception of a single dose of radiation up to 8 Gray (equal to 800 RAD) with palliative intent for pain control up to 14 days before randomization.
* Major surgery within 4 weeks prior to randomization.
* Any known symptomatic brain metastases requiring steroids.
* Women who are pregnant or breastfeeding.
* Gastrointestinal disorder(s) which, in the opinion of the Qualified/Principal Investigator, would significantly impede the absorption of an oral agent (e.g. active Crohn's disease, ulcerative colitis, extensive gastric and small intestine resection).
* Unable or unwilling to swallow BBI608/placebo capsules daily.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, clinically significant non-healing or healing wounds, symptomatic congestive heart failure, unstable angina pectoris, clinically significant cardiac arrhythmia, significant pulmonary disease (shortness of breath at rest or mild exertion), uncontrolled infection or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with a history of other malignancies except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≥ 5 years.
* Prior treatment with BBI608.
* Any active disease condition which would render the protocol treatment dangerous or impair the ability of the patient to receive protocol therapy.
* Any condition (e.g. psychological, geographical, etc.) that does not permit compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2013-05-10 (Actual); Primary Completion 2016-05-07 (Actual); Study Completion 2016-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek Jonker, Study Chair — Ottawa Health Research Institute - General Division
Locations (63):
- Australia (9):
  - Bankstown/ Lidcombe, Bankstown, New South Wales
  - Townsville Hospital, Douglas, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Peter MacCallum Cancer Institute, East Melbourne, Victoria
  - St John of God - Subiaco, Subiaco, Western Australia
  - St John of God Bunbury Hospital, Bunbury
- Canada (39):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Abbotsford Centre, Abbotsford, British Columbia
  - BCCA - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - BCCA - Vancouver Island Cancer Centre, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Horizon Health Network,, Fredericton, New Brunswick
  - The Moncton Hospital, Moncton, New Brunswick
  - The Vitalite Health Network - Dr. Leon Richard, Moncton, New Brunswick
  - Atlantic Health Sciences Corporation, Saint John, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - The Royal Victoria Hospital, Barrie, Ontario
  - Health Sciences North, Greater Sudbury, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Algoma District Cancer Program, Sault Ste. Marie, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Hopital de la Cite-de-la-Sante, Laval, Quebec
  - L'Hotel-Dieu de Levis, Lévis, Quebec
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University - Dept. Oncology, Montreal, Quebec
  - CHUQ-Pavillon Hotel-Dieu de Quebec, Québec, Quebec
  - CHA-Hopital Du St-Sacrement, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - Centre hospitalier regional de Trois-Rivieres, Trois-Rivières, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Japan (15):
  - Chiba Cancer Center, Chiba
  - National Kyushu Cancer Center, Fukuoka
  - National Cancer Center Hospital East, Kashiwa
  - Kobe City Medical Center General Hospital, Kobe
  - National Hospital Organization Shikoku Cancer Center, Matsuyama
  - Kyorin University Hospital, Mitaka
  - Aichi Cancer Center Hospital, Nagoya
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka
  - Saitama Prefectural Cancer Center, Saitama
  - Hokkaido University Hospital, Sapporo
  - Shizuoka Cancer Center, Shizuoka
  - Osaka Medical College Hospital, Takatsuki
  - Cancer Institute Hospital of JFCR, Tokyo
  - Keio University Hospital, Tokyo
  - National Cancer Center Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jonker DJ, Nott L, Yoshino T, Gill S, Shapiro J, Ohtsu A, Zalcberg J, Vickers MM, Wei AC, Gao Y, Tebbutt NC, Markman B, Price T, Esaki T, Koski S, Hitron M, Li W, Li Y, Magoski NM, Li CJ, Simes J, Tu D, O'Callaghan CJ. Napabucasin versus placebo in refractory advanced colorectal cancer: a randomised phase 3 trial. Lancet Gastroenterol Hepatol. 2018 Apr;3(4):263-270. doi: 10.1016/S2468-1253(18)30009-8. Epub 2018 Feb 1. PMID 29397354

RESULTS

PARTICIPANT FLOW:
Groups:
- BBI608: BBI608 480 mg two times daily (960 mg total daily dose)+ Best Supportive Care
  BBI608
  Best Supportive Care
- Placebo: Placebo two times daily + Best Supportive Care
  Placebo
  Best Supportive Care
Period: Overall Study
Arm/Group | BBI608 | Placebo
Started | 138 | 144
Completed | 138 | 144
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients randomized to this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | BBI608 | Placebo | Total
Number analyzed (Participants) | 138 | 144 | 282
Age, Continuous [Median (Full Range); unit: years] | 64 [32 to 85] | 64 [37 to 81] | 64 [32 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 51 | 98
  Male | 91 | 93 | 184
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 26 | 34 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 1 | 1
  White | 112 | 107 | 219
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 64 | 77 | 141
  Japan | 22 | 22 | 44
  Australia | 52 | 45 | 97
ECOG (Eastern Cooperative Oncology Group) Performance Status [Count of Participants; unit: Participants] — 0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    0 | 37 | 42 | 79
    1 | 101 | 102 | 203

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Time from the day of randomization to death. For alive patients, overall survival was censored at the last day the patient was known alive (LKA).
Time Frame: 36 month
Population: All patients who were randomized to this study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BBI608 | Placebo
Number analyzed (Participants) | 138 | 144
Months | 4.44 [3.68 to 4.90] | 4.76 [4.01 to 5.32]
Statistical Analysis 1: Comparison: BBI608 vs Placebo; Test type: Superiority; p = 0.337, Log Rank; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.88 to 1.46]

2. Secondary Outcome: Progression Free Survival
Description: Defined as the time from randomization to the first objective documentation of disease progression or death due to any cause.
Time Frame: 36 months
Population: All patients randomized to this study
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BBI608 | Placebo
Number analyzed (Participants) | 138 | 144
Months | 1.82 [1.74 to 1.87] | 1.82 [1.74 to 1.84]
Statistical Analysis 1: Comparison: BBI608 vs Placebo; Test type: Superiority; p = 0.837, Log Rank; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.76 to 1.26]

3. Secondary Outcome: Disease Control Rate
Description: Proportion of all randomized patients with a documented complete response (CR) defined as disappearance of all target lesions, partial response (PR) defined as >=30% decrease in the sum of the longest diameter of target lesions, and stable disease (SD) defined as <30% decrease but also <20% increase in the sum of the longest diameter of target lesions without new lesions per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) 1.1 for target lesion.
Time Frame: 36 months
Population: All patients randomized to this study
Measure: Count of Participants; unit: Participants
Arm/Group | BBI608 | Placebo
Number analyzed (Participants) | 138 | 144
Participants | 17 | 18
Statistical Analysis 1: Comparison: BBI608 vs Placebo; Test type: Superiority; p = 0.955, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.48 to 2.00]

4. Secondary Outcome: Number of Patients With Adverse Events
Description: Number of patients with at least one adverse event as assessed by NCI CTCAE Version 3.0 criteria.
Time Frame: 36 months
Population: All patients who have received at least one dose of BBI608/Placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | BBI608 | Placebo
Number analyzed (Participants) | 136 | 144
Participants | 135 | 139

5. Secondary Outcome: Change of Global Quality of Life at 8 Weeks From Baseline
Description: Change scores from baseline at time 2 (8 weeks) from baseline for the global health status/quality of life scale scores (between 0 and 100 with higher value indicating better quality of life) as derived from responses of patients to the EORTC (European Organisation for Research and Treatment of Cancer) quality of life questionnaire (QLQ-C30).
Time Frame: 8 weeks
Population: Patients who were assessed Quality of Life at baseline and week 8 from randomization.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BBI608 | Placebo
Number analyzed (Participants) | 55 | 61
units on a scale | -10.61 (23.1) | -10.66 (17.07)
Statistical Analysis 1: Comparison: BBI608 vs Placebo; Test type: Superiority; p = 0.72, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 36 months
Description: Adverse event and/or serious adverse event were collected only from patients who had received at least one dose of protocol treatment. Two patients who were randomized to BBI608 group did not receive any drug and, thus, were not included in the reporting of adverse events.
Groups:
- BBI608: BBI608 480 mg two times daily (960 mg total daily dose)+ Best Supportive Care
  BBI608
  Best Supportive Care
  At risk patients included only patients who received at least one dose of BBI608
- Placebo: Placebo two times daily + Best Supportive Care
  Placebo
  Best Supportive Care
  At risk patients included only patients who received at least one dose of placebo
Arm/Group | BBI608 | Placebo
All-Cause Mortality (participants affected / at risk) | 127/136 | 130/144
Serious Adverse Events (participants affected / at risk) | 40/136 | 29/144
Other Adverse Events (participants affected / at risk) | 134/136 | 137/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BBI608 (N=136) | Placebo (N=144)
Anemia (Blood and lymphatic system disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 0
Bloating (Gastrointestinal disorders) | 0 | 3
Colitis (Gastrointestinal disorders) | 0 | 1
Colonic obstruction (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 6 | 1
Ileal obstruction (Gastrointestinal disorders) | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Jejunal obstruction (Gastrointestinal disorders) | 1 | 2
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 2 | 0
Edema limbs (General disorders) | 0 | 2
Edema trunk (General disorders) | 0 | 1
Fatigue (General disorders) | 2 | 1
Fever (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 2
Non-cardiac chest pain (General disorders) | 1 | 0
Other hepatobiliary disorders (Hepatobiliary disorders) | 1 | 1
Biliary tract infection (Infections and infestations) | 3 | 1
Kidney infection (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 1 | 0
Other infections and infestations (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 2
Upper respiratory infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Intestinal stoma obstruction (Injury, poisoning and procedural complications) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Weight loss (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 7 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Other renal and urinary disorders (Renal and urinary disorders) | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BBI608 (N=136) | Placebo (N=144)
Abdominal pain (Gastrointestinal disorders) | 64 | 56
Bloating (Gastrointestinal disorders) | 8 | 9
Constipation (Gastrointestinal disorders) | 48 | 60
Diarrhea (Gastrointestinal disorders) | 117 | 46
Dry mouth (Gastrointestinal disorders) | 11 | 7
Dyspepsia (Gastrointestinal disorders) | 8 | 17
Gastroesophageal reflux disease (Gastrointestinal disorders) | 10 | 12
Nausea (Gastrointestinal disorders) | 85 | 67
Other gastrointestinal disorders (Gastrointestinal disorders) | 5 | 11
Vomiting (Gastrointestinal disorders) | 60 | 50
Edema limbs (General disorders) | 20 | 29
Fatigue (General disorders) | 92 | 94
Fever (General disorders) | 12 | 15
Pain (General disorders) | 23 | 15
Weight loss (Investigations) | 19 | 11
Anorexia (Metabolism and nutrition disorders) | 76 | 66
Dehydration (Metabolism and nutrition disorders) | 9 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 13
Arthritis (Musculoskeletal and connective tissue disorders) | 7 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 31 | 38
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 14
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 15
Dizziness (Nervous system disorders) | 8 | 13
Dysgeusia (Nervous system disorders) | 8 | 12
Headache (Nervous system disorders) | 15 | 18
Peripheral sensory neuropathy (Nervous system disorders) | 43 | 38
Anxiety (Psychiatric disorders) | 16 | 12
Depression (Psychiatric disorders) | 12 | 8
Insomnia (Psychiatric disorders) | 32 | 34
Urinary frequency (Renal and urinary disorders) | 7 | 5
Urine discoloration (Renal and urinary disorders) | 38 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 34 | 31
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 36 | 45
Dry skin (Skin and subcutaneous tissue disorders) | 9 | 11
Other skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 8 | 9
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 8 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 9
Rash acneiform (Skin and subcutaneous tissue disorders) | 8 | 7
Hypertension (Vascular disorders) | 27 | 24
Thromboembolic event (Vascular disorders) | 9 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No